CLINICAL TRIAL: NCT02105077
Title: Development of a Mass-spectometry Based Method for Detecting Xenon Application in Humans
Status: Completed | Type: Observational
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Collaborators: German Sport University, Cologne (Other)
Responsible Party: Principal Investigator, Klinik für Anästhesiologie, Prof. Dr. Peter Kienbaum, Heinrich-Heine University, Duesseldorf
Other Study IDs: 2014032273
Record Dates: First submitted 2014-03-31; First posted 2014-04-07 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Anesthesia
Keywords: xenon; doping; anesthesia; mass spectrometry; surgery
MeSH Terms: interventions — Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole-blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Xenon: Patients undergoing surgery with xenon-based general anesthesia
  Interventions: Drug: Anesthesia with inhalative application of xenon gas

INTERVENTIONS:
Drug: Anesthesia with inhalative application of xenon gas

SUMMARY:
The purpose of this study is to establish a laboratory method to determine from blood samples whether a person has been treated with xenon.

DETAILED DESCRIPTION:
The noble gas xenon is used for general anesthesia in clinical routine. Recent reports indicate that xenon is also used for increasing performance in high-performance sports. The purpose of this study is to establish a method for detecting xenon exposure in humans.

In patients undergoing surgery with xenon anesthesia as part of routine hospital care, small blood samples (3ml) will be taken before anesthesia, during anaesthesia and at 1,2, 4, 8, 16, 24, 32, 40 and 48 hours after anesthesia. These blood samples will be analyzed for traces of xenon.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years and older
* Xenon-based anesthesia as part of routine care

Exclusion Criteria:

* Inability to give written informed consent
* Known pregnancy
* Hemoglobin concentration of less than 12g/dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing xenon-based general anesthesia as part of routine care at University Hospital Düsseldorf, Germany
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2014-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Detection of xenon in patient blood sample by mass spectrometry | Immediately before induction of anesthesia
Detection of xenon in patient blood sample by mass spectrometry | During xenon anesthesia
Detection of xenon in patient blood sample by mass spectrometry | 4 hours after extubation
Detection of xenon in patient blood sample by mass spectrometry | 8 hours after extubation
Detection of xenon in patient blood sample by mass spectrometry | 24 hours after xenon anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Klinik für Anästhesiologie, Universitätsklinikum Düsseldorf, Düsseldorf, Germany